CLINICAL TRIAL: NCT06543329
Title: Comparative Analysis Between Different Suture Materials in Subcuticular Cesarean Wound Closure in Woman With BMI 40 or Greater in Cesarean Delivery: An Interventional Randomized Comparative Clinical Trial
Brief Title: Comparative Analysis of Subcuticular Suture Materials in Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AA-2024-3
Record Dates: First submitted 2024-07-27; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cesarean Wound Disruption With Postnatal Complication
Keywords: cesarean section; wound complication; obesity; monocryl; vicryl; prolene; polyester
MeSH Terms: conditions — Obesity | interventions — Polyglactin 910; glycolide E-caprolactone copolymer; Polypropylenes; Polyesters

STUDY DESIGN:
Intervention Model Description: This prospective interventional randomized comparative clinical trial was carried out on 300 pregnant women scheduled for elective caesarean section at operative theater
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- polyglactin 910 (Active Comparator): - Group A: (75) women with subcuticular suture polyglactin 910, braided, (VICRYL RAPIDE®; Ethicon) was used in subcuticular skin closure.
  Interventions: Procedure: polyglactin 910
- poliglecaprone 25 (Active Comparator): Group A: (75) women with subcuticular suture poliglecaprone 25, (MONOCRYL) was used in subcuticular skin closure.
  Interventions: Procedure: poliglecaprone 25
- polypropylene (Active Comparator): Group A: (75) women with subcuticular suture polypropylene, (PROLENE) was used in subcuticular skin closure.
  Interventions: Procedure: polypropylene
- POLYESTER (Active Comparator): Group A: (75) women with subcuticular suture POLYESTER, (ETHIBOND EXCEL Suture) was used in subcuticular skin closure.
  Interventions: Procedure: polyester

INTERVENTIONS:
Procedure: polyglactin 910 — 75 PARTICIPANT, Vicryl suture was used in subcuticular suture
  Other Names: VICRYL
  Arms: polyglactin 910
Procedure: poliglecaprone 25 — 75 PARTICIPANT, monocryl suture was used in subcuticular suture
  Other Names: monocryl
  Arms: poliglecaprone 25
Procedure: polypropylene — 75 PARTICIPANT, Prolene suture was used in subcuticular suture
  Other Names: prolene
  Arms: polypropylene
Procedure: polyester — 75 PARTICIPANT, Polyester suture was used in subcuticular suture
  Other Names: ETHIBOND EXCEL Suture
  Arms: POLYESTER

SUMMARY:
1.1. Background and Rationale Cesarean section is one of the most common surgical procedures performed worldwide. The choice of suture material for closing the skin incision is crucial, as it can influence wound healing, the risk of wound complications, and the cosmetic outcome. Subcuticular suturing, a technique where the suture is placed just under the skin, is favored for its aesthetic benefits and reduced risk of infection. However, the type of suture material used can significantly impact these outcomes. This study aims to provide a comparative analysis of various subcuticular suture materials used in cesarean sections, focusing on wound complications and incision outcomes.

1.2. Objective of the Study The objective of this study is to compare the incidence of wound complications and the quality of incision outcomes associated with different subcuticular suture materials used in cesarean sections. By doing so, the investigators aim to identify the most effective suture material for minimizing wound complications and optimizing cosmetic results.

DETAILED DESCRIPTION:
2.1. Surgical Techniques in Cesarean Section Cesarean section involves multiple surgical steps, including skin incision, uterine incision, and closure of the incisions. The subcuticular suturing technique is often preferred for skin closure due to its potential for better cosmetic results and lower infection rates compared to other methods like staples or interrupted sutures.

2.2. Types of Suture Materials

Suture materials can be broadly categorized into absorbable and non-absorbable, and further into monofilament and multifilament types. Common suture materials used in subcuticular skin closure include:

Absorbable Sutures: Poliglecaprone (Monocryl), Polyglactin (Vicryl), Polydioxanone (PDS).

Non-Absorbable Sutures: Nylon, Polypropylene (Prolene), Silk. 2.3. Previous Studies on Suture Materials in Cesarean Section Previous studies have explored the impact of different suture materials on wound healing, infection rates, and cosmetic outcomes. Research indicates varying results, with some studies favoring absorbable sutures for their reduced need for removal and lower infection rates, while others suggest non-absorbable sutures may provide stronger wound support. However, comprehensive comparative analyses specific to cesarean sections remain limited.

3. Methodology 3.1. Study Design This study will use a prospective, randomized controlled trial design. Participants undergoing elective cesarean sections will be randomly assigned to receive subcuticular suturing with one of several suture materials.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20-45 years old.
2. BMI = or more than 40 kg/m2
3. Primigravida or not more than the previous 1 cesarean section.
4. Will undergo a lower-segment cesarean section.
5. Hb: ≥ 10 gm/dl.
6. Viable fetus.
7. No history of medical comorbidities.

Exclusion Criteria:

1. History of urogenital tract infection within 2 weeks before cesarean delivery.
2. Presence of clinical signs of infection at the time of delivery including PPROM and intraamniotic infection.
3. Medical comorbidities (hypertension, diabetes, etc.).
4. Hypersensitivity to any of the suture materials.
5. Women with abnormal placentation (placental abruption or placenta previa).
6. History of systemic corticosteroid intake during their pregnancy for 2 weeks or more.
7. History of previous surgical site infection.
8. Immune-compromised women.
9. Women refused to participate in the study or could not obtain consent.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This prospective interventional randomized comparative clinical trial was carried out on 300 pregnant women scheduled for elective caesarean section at operative theater
Enrollment: 300 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
the rate of any documented wound complication during the first six weeks postpartum | 6 weeks
  This measure tracks the incidence of wound complications within six weeks postpartum, including infection, dehiscence, seroma, hematoma, ecchymosis, pus, delayed healing, and secondary suture needs.
  Measurement Tools:
  Clinical examinations during follow-up visits Patient self-reports Review of medical records
  Assessment Procedure:
  Patients will undergo follow-up visits at 2, 4, and 6 weeks postpartum. Complications will be documented through clinical exams, patient reports, and medical record reviews.
  Calculation:
  The rate is calculated as the number of patients with any wound complication divided by the total number of patients, expressed as a percentage.

SECONDARY OUTCOMES:
cosmetics satisfaction | 6 weeks
  This measure assesses the cosmetic appearance of surgical wounds post-abdominal myomectomy.
  Measurement Tool:
  A standardized cosmetic appearance scale will be used, such as the Patient and Observer Scar Assessment Scale (POSAS).
  Assessment Procedure:
  Evaluations will be conducted at follow-up visits (2, 4, and 6 weeks postpartum) by both the patient and a clinician.
  Parameters Assessed:
  Scar color, texture, and overall appearance Patient satisfaction with the cosmetic outcome
  Calculation:
  Scores from the POSAS will be averaged to determine the overall cosmetic appearance rating.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed N Afifi, MD, Principal Investigator — Kafrelsheikh University
Locations (1):
- faculty of medicine, Kasr el ainy hospital, Cairo university, Cairo, Egypt

REFERENCES:
- [Background] Rodel RL, Gray KM, Quiner TE, Bodea Braescu A, Gerkin R, Perlow JH. Cesarean wound closure in body mass index 40 or greater comparing suture to staples: a randomized clinical trial. Am J Obstet Gynecol MFM. 2021 Jan;3(1):100271. doi: 10.1016/j.ajogmf.2020.100271. Epub 2020 Oct 27. PMID 33451603
- [Background] Basha SL, Rochon ML, Quinones JN, Coassolo KM, Rust OA, Smulian JC. Randomized controlled trial of wound complication rates of subcuticular suture vs staples for skin closure at cesarean delivery. Am J Obstet Gynecol. 2010 Sep;203(3):285.e1-8. doi: 10.1016/j.ajog.2010.07.011. PMID 20816153
- [Background] Frishman GN, Schwartz T, Hogan JW. Closure of Pfannenstiel skin incisions. Staples vs. subcuticular suture. J Reprod Med. 1997 Oct;42(10):627-30. PMID 9350017
- [Background] Clay FS, Walsh CA, Walsh SR. Staples vs subcuticular sutures for skin closure at cesarean delivery: a metaanalysis of randomized controlled trials. Am J Obstet Gynecol. 2011 May;204(5):378-83. doi: 10.1016/j.ajog.2010.11.018. Epub 2010 Dec 31. PMID 21195384
- [Background] Tuuli MG, Rampersad RM, Carbone JF, Stamilio D, Macones GA, Odibo AO. Staples compared with subcuticular suture for skin closure after cesarean delivery: a systematic review and meta-analysis. Obstet Gynecol. 2011 Mar;117(3):682-690. doi: 10.1097/AOG.0b013e31820ad61e. PMID 21343772
- [Background] Nayak G B, Saha PK, Bagga R, Joshi B, Rohilla M, Gainder S, Sikka P. Wound complication among different skin closure techniques in the emergency cesarean section: a randomized control trial. Obstet Gynecol Sci. 2020 Jan;63(1):27-34. doi: 10.5468/ogs.2020.63.1.27. Epub 2019 Dec 23. PMID 31970125
- [Background] Aabakke AJM, Krebs L, Pipper CB, Secher NJ. Subcuticular suture compared with staples for skin closure after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2013 Oct;122(4):878-884. doi: 10.1097/AOG.0b013e3182a5f0c3. PMID 24084548
- [Background] Buresch AM, Van Arsdale A, Ferzli M, Sahasrabudhe N, Sun M, Bernstein J, Bernstein PS, Ngai IM, Garry DJ. Comparison of Subcuticular Suture Type for Skin Closure After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2017 Sep;130(3):521-526. doi: 10.1097/AOG.0000000000002200. PMID 28796687
- [Background] Figueroa D, Jauk VC, Szychowski JM, Garner R, Biggio JR, Andrews WW, Hauth J, Tita AT. Surgical staples compared with subcuticular suture for skin closure after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2013 Jan;121(1):33-8. doi: 10.1097/aog.0b013e31827a072c. PMID 23262925